CLINICAL TRIAL: NCT07323797
Title: Overlapping Pelvic and Temporomandibular Pain: A Cross-Sectional Analysis of Psychosocial and Sensitization Mechanisms
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Associate Professor, University of Valencia
Other Study IDs: 2025-FIS-4199837
Record Dates: First submitted 2025-12-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pain
Keywords: Chronic Pain; Comorbidity; Cross-sectional; Pelvic Pain; Temporomandibular Joint Disorders
MeSH Terms: conditions — Pain; Chronic Pain; Pelvic Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chronic Pain: Adults with chronic pain who do not report pain in the pelvic region or the temporomandibular joint.
- Temporomandibular Pain Only: Adults with chronic pain who report pain or dysfunction in the temporomandibular joint region but do not report pelvic pain.
- Pelvic Pain Only: Adults with chronic pain who report pelvic pain but do not report temporomandibular joint pain.
- Overlapping Pelvic and Temporomandibular Pain: Adults with chronic pain who report both pelvic pain and temporomandibular joint pain, consistent with chronic overlapping pain conditions.

SUMMARY:
The goal of this observational study is to learn whether pain in the temporomandibular joint is associated with pelvic pain in adults, and to explore psychosocial and pain sensitization factors that may contribute to both conditions.

The main questions it aims to answer are:

Is temporomandibular joint dysfunction associated with pelvic pain in the adult population? Are psychosocial factors and indicators of central pain sensitization related to the co-occurrence of these pain conditions?

Participants will complete standardized, self-administered questionnaires at a single point in time that assess:

Temporomandibular joint symptoms Pelvic pain symptoms Psychosocial factors and pain sensitization features

No treatments or interventions will be given as part of this study.

DETAILED DESCRIPTION:
Chronic pain is a major public health concern due to its high prevalence and its significant impact on quality of life, daily functioning, and overall well-being. Among chronic pain types, nociplastic pain is characterized by persistent pain in the absence of clear tissue damage and is associated with alterations in central pain processing, including central sensitization and dysfunction of the central nervous system. These alterations may manifest as widespread pain sensitivity, autonomic dysregulation, and changes in sensory integration, contributing to long-lasting and diffuse pain experiences.

Individuals with chronic pain frequently report pain in more than one body region, a phenomenon known as Chronic Overlapping Pain Conditions (COPC). The presence of overlapping pain conditions suggests shared underlying mechanisms, such as central sensitization and common psychosocial modulators, which may explain the co-occurrence of different chronic pain syndromes. In this context, temporomandibular joint (TMJ) pain and pelvic pain are of particular interest, as emerging evidence indicates a possible association between these conditions.

Given the existing evidence linking chronic pain conditions across different body regions, further investigation into the co-occurrence of TMJ dysfunction and pelvic pain is warranted. This observational, cross-sectional study aims to characterize the association between these two pain conditions in an adult population and to explore demographic, socioeconomic, psychosocial, and pain-related factors that may help explain their relationship. By improving understanding of shared pain mechanisms, this research seeks to inform future clinical approaches that are more comprehensive and integrative.

Data will be collected at a single time point using standardized, self-administered questionnaires, in accordance with the STROBE guidelines for observational research. Demographic variables will include age, sex, and-among female participants-reproductive and hormonal history (pregnancy, childbirth, episiotomy, cesarean section, and menopausal status). Additional variables will include marital status, current medication use, height, weight, smoking status, physical activity levels, and the duration of orofacial and/or pelvic pain symptoms. Socioeconomic factors such as educational level, classified according to the International Standard Classification of Education (ISCED), and monthly household income, categorized into national income deciles, will also be recorded.

The co-occurrence of chronic pain conditions will be assessed using the Chronic Overlapping Pain Conditions Screener (COPC-S). Pain intensity will be measured using the Numerical Rating Scale (NRS), while fear of movement related to orofacial pain will be evaluated using the Tampa Scale of Kinesiophobia adapted for temporomandibular disorders (TSK-TMD). The presence of central sensitization symptoms will be assessed with the Central Sensitization Inventory (CSI). Psychosocial influences on pain will be examined through measures of health-related quality of life (Short Form-12), perceived stress (Perceived Stress Scale-10), and anxiety (short form of the State-Trait Anxiety Inventory, STAI-6).

By systematically examining the overlap between temporomandibular and pelvic pain and their associated biopsychosocial factors, this study aims to provide preliminary evidence on shared mechanisms of chronic pain. The findings may support the development of more holistic assessment strategies and integrated clinical interventions for individuals experiencing chronic overlapping pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Presence of chronic pain
* Ability to complete self-administered questionnaires.
* Signed informed consent provided prior to participation.

Exclusion Criteria:

* Inability to read or understand Spanish.
* Failure or refusal to provide informed consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from the adult general population experiencing chronic pain. The study population includes individuals aged 18 years or older who report pain in the orofacial (temporomandibular) region, the pelvic region, both regions, or chronic pain in other body areas without involvement of the temporomandibular or pelvic regions. Participants must be able to read and understand Spanish and provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Co-occurrence of Chronic Pain Conditions | Baseline
  The presence and degree of overlapping chronic pain conditions will be assessed using the Chronic Overlapping Pain Conditions Screener (COPC-S). This validated tool identifies co-occurring pain conditions across different body regions and will be used to classify participants into pain groups and to quantify overlap between temporomandibular and pelvic pain.

SECONDARY OUTCOMES:
Pain Intensity | Baseline
  Pain intensity in the temporomandibular and/or pelvic regions will be measured using the Numerical Rating Scale (NRS). Participants will rate their pain intensity on an 11-point scale ranging from 0 (no pain) to 10 (worst pain imaginable). The NRS is a widely used and validated measure of pain severity in chronic pain populations.
Kinesiophobia Related to Temporomandibular Pain | Baseline
  Fear of movement related to orofacial pain will be assessed using the Tampa Scale of Kinesiophobia for Temporomandibular Disorders (TSK-TMD), a validated and culturally adapted version of the original Tampa Scale of Kinesiophobia. The TSK-TMD is a self-reported questionnaire that evaluates pain-related fear and avoidance behaviors associated with jaw movement in individuals with temporomandibular disorders. Total scores range from 17 to 68, with higher scores indicating greater levels of kinesiophobia (worse outcome).
Central Sensitization Symptoms | Baseline
  Central sensitization-related symptoms will be assessed using the Central Sensitization Inventory (CSI), Spanish-validated version. The CSI is a self-reported questionnaire designed to evaluate symptoms associated with altered central pain processing, including widespread pain, fatigue, sleep disturbances, and cognitive difficulties. The total score ranges from 0 to 100, with higher scores indicating a greater severity of central sensitization symptoms (worse outcome).
Health-Related Quality of Life | Baseline
  Health-related quality of life will be assessed using the Short Form-12 Health Survey (SF-12), Spanish-validated version. The SF-12 is a self-reported instrument that generates two composite scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS), reflecting physical and mental aspects of overall functioning and well-being. Each composite score is standardized to range from 0 to 100, with higher scores indicating better perceived health status (better outcome).
Perceived Stress | Baseline
  Perceived stress levels will be assessed using the Perceived Stress Scale-10 (PSS-10), a self-reported questionnaire that evaluates the degree to which individuals perceive their lives as stressful during the past month. The total score ranges from 0 to 40, with higher scores indicating greater perceived stress (worse outcome).
Anxiety Levels | Baseline
  Anxiety will be assessed using the State-Trait Anxiety Inventory, 6-item short form (STAI-6), a self-reported instrument designed to measure current (state) anxiety symptoms and emotional tension. Total scores range from 6 to 24, with higher scores indicating greater anxiety levels (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No